CLINICAL TRIAL: NCT02814461
Title: A Phase I Clinical Trial Evaluating the Safety and Maximum Tolerated Dose of Axitinib in Combination With Radiotherapy for Advanced Hepatocellular Carcinoma (HCC)
Brief Title: The Safety and Maximum Tolerated Dose of Axitinib in Combination With Radiotherapy for HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150704M
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Axitinib; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental): Combined axitinib and radiotherapy (fixed strength)
  Interventions: Drug: Axitinib; Radiation: Radiation

INTERVENTIONS:
Drug: Axitinib — Axitinib (dose escalation): for total 8 weeks during and after RT, with starting dose of 1mg BID. According to the rule of traditional 3 + 3 design, 3-level axitinib dose escalation will be conducted: 1mg BID (level - I), 2mg BID (level - II) and 3mg BID (level - III).
  Other Names: Inlyta
Radiation: Radiation — Radiotherapy (RT) dose (fixed strength for normal liver): 37.5 to 67.5 Gy in 15 fractions (2.5 to 4.5 Gy per fraction) to liver tumor(s) (e.g. portal vein thrombosis, tumors with size ≥3 cm, or recurrent/refractory tumors). The final prescribed dose is based on an upper limit of mean liver dose of 18 Gy for all plans. (Daily Entecavir 0.5-1mg or Telbivudine 600mg is recommended for patients with positive hepatitis B during and 3 months after RT.)

SUMMARY:
To determine the maximal tolerated dose (MTD) of axitinib in combination with RT for advanced HCC.

DETAILED DESCRIPTION:
The goal of this study is to conduct a phase I clinical trial evaluating the safety and MTD of axitinib in combination with RT for advanced HCC. There are some rationales of conducting this clinical trial. Firstly, there is evidence of benefit from the combination of a variety of anti-angiogenic agents with RT at the pre-clinical level. Numerous pre-clinical models have documented improved outcome with the combination of RT (e.g. bevacizumab ... etc). Potential increasing the oxygenation of tumors with anti-angiogenesis is also expected to improve the therapeutic ratio of radiation therapy to hypervascular caner like HCC. Secondly, spatial cooperation may exist between local treatment (e.g. RT) and systemic therapy (e.g. axitinib). From the experience of sorafenib, the majority of patients eventually progress within the liver and die of liver failure, providing rationale to use local therapies like RT. On the other hand, from the experience of RT, the most common site of first recurrence was in the liver outside the irradiated volume, providing rationale for studies combining regional or systemic therapies with RT. Thirdly, clinical experiences with RT and anti-angiogenic agent are few but still exist with encouraging results. For example, one retrospective review from Taiwan with advanced HCC treated with RT and sunitinib (a TKI with similar mechanisms as sorafenib) reported objective response rate of 74% and a median survival of 16 months, and concluded hypofractionated RT and sunitinib can be delivered safely in HCC patients, which was compatible with the result of several phase I or II studies using sorafenib plus. Fourthly, the safety and MTD of axitinib combined with RT is needed to be established before launch of a phase II study

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-85 years, with ECOG performance 0-2.
* Advanced hepatocellular carcinoma (HCC), histologically or clinically diagnosed. (Multiple tumors, portal vein thrombosis, nodal metastasis or distant metastasis is allowed.)
* Unsuitable for resection, liver transplantation, radiofrequency ablation (RFA) or transarterial chemoembolization (TACE), or recurrent / refractory after prior local-regional treatment.
* ≥ One measurable tumor.
* Child-Pugh score A or B.
* Patients who fulfill all of the following criteria:

  1. Serum total bilirubin ≤ 3 mg/dL
  2. Serum alanine transaminase (ALT) ≤ 5 times ULN
  3. INR ≤ 2.20
  4. Platelet count ≥ 50,000 /mm3
  5. WBC count ≥ 3,000 /mm3 or ANC ≥ 1,500 /mm3
  6. Serum creatinine ≤ 2.0 mg/dL
* Normal thyroid function confirmed.
* Absence of grant for sorafenib.
* Sorafenib failure or intolerability (if ever used).

Exclusion Criteria:

* Considered to have high risk of bleeding (e.g. active peptic ulcer, unstable esophageal/gastric varices, history of aneurysm, and requirement of anticoagulant therapy).
* Pre-existing uncontrolled hypertension (systolic >140 mmHg, diastolic >90 mmHg) or proteinuria ≧500 mg/24 hours.
* Prior history of coronary artery disease.
* The patient is participating in other clinical trials.
* Pregnant women.
* Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Patients with non-healing wound.
* Requiring the use of potent CYP3A4/5 inhibitors or inducers (see Appendix).
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The maximal tolerated dose (MTD) | Within 12 weeks
  To determine the maximal tolerated dose (MTD) of axitinib in combination with RT for advanced HCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang KL, Chi MS, Ko HL, Huang YY, Huang SC, Lin YM, Chi KH. Axitinib in combination with radiotherapy for advanced hepatocellular carcinoma: a phase I clinical trial. Radiat Oncol. 2021 Jan 20;16(1):18. doi: 10.1186/s13014-020-01742-w. PMID 33472666